CLINICAL TRIAL: NCT03816241
Title: Mechanisms of Nudges on Families' Decision-Making Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSS-1502-P02-05
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Organ Donation
MeSH Terms: interventions — Reading Frames

STUDY DESIGN:
Intervention Model Description: Participants are assigned to 1 out of 4 possible anecdotes; Control, Framing, Norms, Combination.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Vignette contains no extra information.
- Frame (Experimental): Vignette is framed in a particular manner
  Interventions: Other: Frame
- Norms (Experimental): Vignette contains extra information about norms
  Interventions: Other: Norms
- All (Experimental): Vignette contains extra information about norms and is framed in a particular manner.
  Interventions: Other: Frame; Other: Norms

INTERVENTIONS:
Other: Frame — Vignette is framed in a way that nudges participant to leave a legacy
  Arms: All; Frame
Other: Norms — Vignette informs the participant that most people choose an option to try to nudge participant into choosing that option as well
  Arms: All; Norms

SUMMARY:
As part of a larger study, participants are told to read 1 out of 4 anecdotes depicting an organ donation scenario where they are required to make a decision on behalf of their mother who has just suffered an accident. The participants are then surveyed on their attitudes towards organ donation.

DETAILED DESCRIPTION:
As part of a larger study, participants are given 1 out of 4 possible vignettes which depicts an organ donation scenario involving their mother. The possible vignettes consist of a Control condition, a Framing condition, a Normative condition and a condition that includes all the nudges. Participants are then given surveys to gauge their views and attitudes towards organ donation as a whole, their trust towards medical institutions and the doctors, their perceived manipulation from the doctor and their views on the altruistic nature of organ donation.

ELIGIBILITY:
Inclusion Criteria:

* Above age 21
* Singapore Citizens and Permanent Residents

Exclusion Criteria:

* Below age 21
* Non-citizens
* Not able to make decisions for self

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
5-point Likert scale - Trust and Perceived Manipulativeness of doctor and medical institution | 3 minutes
  A 5-point Likert scale will be given and participants will be asked to rate their agreeableness towards the level of trust and perceived manipulativeness of the doctor and the medical institution.
9-point rating scale - Views on altruistic nature of organ donation | 1 minute
  A 9-point rating scale will be given and participants will be asked to rate their views on the meaningfulness of organ donation.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided